CLINICAL TRIAL: NCT00917150
Title: A Phase 2, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-arm, Dose-comparison Trial of OPC-6535 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: To Investigate the Efficacy and Safety of OPC-6535 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 197-08-801; JapicCTI-090770
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — tetomilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- OPC-6535 12.5mg (Experimental)
  Interventions: Drug: tetomilast (OPC-6535)
- OPC-6535 25mg (Experimental)
  Interventions: Drug: tetomilast (OPC-6535)
- OPC-6535 50mg (Experimental)
  Interventions: Drug: tetomilast (OPC-6535)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tetomilast (OPC-6535) — oral administration of 12.5mg OPC-6535, once daily for 24months
  Arms: OPC-6535 12.5mg
Drug: tetomilast (OPC-6535) — oral administration of 25mg OPC-6535, once daily for 24months
  Arms: OPC-6535 25mg
Drug: tetomilast (OPC-6535) — oral administration of 50 mg OPC-6535, once daily for 24months
  Arms: OPC-6535 50mg
Drug: placebo — oral administration of placebo, once daily for 24months
  Arms: placebo

SUMMARY:
To investigate the efficacy and safety of OPC-6535 in COPD patients, using the measurement of trough FEV1 over time as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years, inclusive, at the time informed consent is obtained
* Ability to provide own written informed consent
* Agree to use an appropriate method of contraception until 3 months after the last dose of the investigational medicinal product (IMP)
* A rating of 1 or higher on the Goddard scale in assessment of emphysema severity by chest CT scan at screening
* Ratio of forced expiratory volume in 1 second to forced vital capacity (FEV1/FVC) of less than 70% at screening
* Cigarette smoking history of at least 20 pack years at screening

Exclusion Criteria:

* Subjects with obstructive disorders due to bronchial asthma
* Subjects receiving long-term oxygen therapy
* Subjects with active tuberculosis or obvious bronchiectasis
* Complication of malignant tumor
* Uncontrolled cardiovascular, endocrine, blood, or nervous system disorders
* Uncontrolled condition with COPD exacerbation of level 2 or 3 within 8 weeks prior to the start of washout period (within 12 weeks prior to start of treatment period)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2009-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- China (7):
  - Central China Area
  - East China Area
  - North China Area
  - Northeast China Area
  - Northwest China Area
  - South China Area
  - Southwest China Area
- Kansai Region, Et Al., Japan
- Seoul, Et Al., South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-6535 12.5 mg: Oral administration of 12.5mg OPC-6535 once daily for 24 months
- OPC-6535 25 mg: Oral administration of 25mg OPC-6535 once daily for 24 months
- OPC-6535 50 mg: Oral administration of 50 mg OPC-6535 once daily for 24 months (started from 25 mg for the first 2 weeks and the dose was titrated to 50 mg from the third week)
- Placebo: Oral administration of placebo once daily for 24 months
Period: Overall Study
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Started | 192 | 198 | 191 | 190
Completed | 155 | 161 | 149 | 156
Not Completed | 37 | 37 | 42 | 34
Not completed — Adverse Event | 12 | 7 | 12 | 11
Not completed — Death | 1 | 4 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 4 | 2
Not completed — Physician Decision | 0 | 2 | 0 | 1
Not completed — Protocol Violation | 5 | 5 | 3 | 5
Not completed — Withdrawal by Subject | 15 | 16 | 18 | 11
Not completed — Other than specified | 3 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted all subjects randomized to double-blind therapy, regardless of any protocol violation.
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo | Total
Number analyzed (Participants) | 192 | 198 | 191 | 190 | 771
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (7.63) | 64.0 (7.01) | 63.2 (7.55) | 63.4 (7.24) | 63.2 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 18 | 15 | 54
  Male | 178 | 191 | 173 | 175 | 717
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 32 | 37 | 35 | 32 | 136
  Japan | 12 | 13 | 10 | 10 | 45
  China | 148 | 148 | 146 | 148 | 590

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) Change From Baseline to 24 Months
Description: Measurement over time (from baseline over the 24-month treatment period) and change from baseline to end of the treatment period.
Time Frame: Baseline, 24 months
Population: ITT population consisted of all subjects randomized to double-blind therapy, regardless of any protocol violation.
Measure: Mean (Standard Error); unit: Liters
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 152 | 163 | 152 | 149
Liters | -0.004 (0.0481) | -0.023 (0.0481) | -0.018 (0.0473) | -0.035 (0.0480)

2. Secondary Outcome: Change From Baseline at 24 Months in Total Symptom Diary Score
Description: Subjects were required to keep a symptom diary throughout the entire trial period from the start of investigational medicinal product (IMP) administration in the washout period until the end of the treatment period. Assessment items included scores for shortness of breath, cough, and sputum, IMP compliance, use of salbutamol and respiratory symptom medications, and smoking status. Subjects recorded a score of between 0 and 3, with 0 indicating no symptoms and 3 indicating a high level of symptoms, for each domain.
Time Frame: Baseline, 24 months
Population: ITT population consisted of all subjects randomized to double-blind therapy, regardless of any protocol violation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 150 | 161 | 152 | 151
score on a scale | 0.063 (0.0606) | 0.073 (0.0606) | 0.077 (0.0597) | 0.101 (0.0606)

3. Secondary Outcome: Change From Baseline at 24 Months in St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ is a self-administered questionnaire designed to measure and quantify the impact of chronic respiratory disease on health-related quality of life (QOL) and well-being in three domains: symptoms, activity, and impact on daily life. The SGRQ was completed by each subject prior to IMP administration at baseline and at Month 6, Month 12, Month 18, and Month 24 (end of treatment).
  A weighted score based on population norms for each dimension and total was evaluated. Scores were expressed as a percentage of overall impairment where 100 represented worst possible health status and 0 indicated best possible health status. Scores were calculated when less than 24% of the item scores were missing, otherwise the scores were set to missing. Where there were multiple answers for a question, the worst case was used.
Time Frame: Baseline, 24 months
Population: ITT population consisted of all subjects randomized to double-blind therapy, regardless of any protocol violation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 151 | 157 | 148 | 151
score on a scale | -9.6 (3.80) | -7.9 (3.80) | -7.7 (3.73) | -10.4 (3.80)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the start of IMP administration until follow-up (2 weeks after the end of treatment or early termination)
Description: Safety analyses were conducted on the safety population, defined all randomized subjects who took at least one dose of the IMP. A TEAE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the IMP, regardless of judgment of relationship to the IMP.
Arm/Group | OPC-6535 12.5 mg | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/192 | 5/196 | 3/191 | 2/190
Serious Adverse Events (participants affected / at risk) | 47/192 | 47/196 | 50/191 | 46/190
Other Adverse Events (participants affected / at risk) | 108/192 | 116/196 | 102/191 | 105/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 12.5 mg (N=192) | OPC-6535 25 mg (N=196) | OPC-6535 50 mg (N=191) | Placebo (N=190)
Chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 22 | 24 | 22 | 24
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 2 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster infection neurological (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary tuberculoma (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Large cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Colonic polyp (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 1 | 2 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cor pulmonale chronic (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hypoxic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal meningeal cyst (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Computerised tomogram thorax abnormal (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Chronic granulomatous disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyssomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 12.5 mg (N=192) | OPC-6535 25 mg (N=196) | OPC-6535 50 mg (N=191) | Placebo (N=190)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 58 | 67 | 52 | 57
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 2 | 3
Nasopharyngitis (Infections and infestations) | 33 | 21 | 19 | 22
Pneumonia (Infections and infestations) | 4 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 18 | 8
Abdominal pain upper (Gastrointestinal disorders) | 8 | 11 | 10 | 3
Gastritis (Gastrointestinal disorders) | 3 | 7 | 9 | 5
Abdominal distension (Gastrointestinal disorders) | 4 | 4 | 6 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3 | 8 | 1
Toothache (Gastrointestinal disorders) | 4 | 4 | 2 | 3
Nausea (Gastrointestinal disorders) | 3 | 2 | 5 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 5 | 2 | 5 | 4
Protein urine present (Investigations) | 1 | 4 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 3 | 3
Headache (Nervous system disorders) | 7 | 8 | 3 | 3
Dizziness (Nervous system disorders) | 2 | 7 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | 10 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 2 | 4 | 1
Pyrexia (General disorders) | 4 | 3 | 5 | 1
Proteinuria (Renal and urinary disorders) | 5 | 2 | 2 | 3
Hypertension (Vascular disorders) | 4 | 8 | 5 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 | 4 | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 4 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No